CLINICAL TRIAL: NCT06716801
Title: Observational Cohort Study on Adult Patients With Not-adequately Controlled FOcal-onset Seizures Treated With Cenobamate as Early adjUnctive Therapy in a Real-world Setting - FOCUS
Brief Title: Real-world Clinical Response to Cenobamate Early add-on in France, Germany and Spain
Status: Recruiting | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 169(A)MD23324
Record Dates: First submitted 2024-11-22; First posted 2024-12-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-11

CONDITIONS: Focal Epilepsy With and Without Secondary Generalization
Keywords: focal-onset seizures; epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Cenobamate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by epilepsy with focal-onset seizures with or without secondary generalization: Adult patients affected by epilepsy with focal-onset seizures with or without secondary generalization who have not been adequately controlled despite a history of treatment with 2 or 3 anti-seizure medications (ASMs).
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — Adult patients affected by epilepsy with focal-onset seizures with or without secondary generalization who have not been adequately controlled despite a history of treatment with 2 or 3 anti-seizure medications.

SUMMARY:
Aim of the study is to better characterize the clinical profile of adjunctive cenobamate by collecting data from the current standard clinical practice in France, Germany, and Spain, to describe the real-world clinical response among adult patients affected by focal epilepsy not adequately controlled despite a history of 2 or 3 ASMs before starting treatment with cenobamate (including previous and concomitant ASMs).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years old at the time of cenobamate treatment initiation.
2. Patients with a diagnosis of epilepsy with focal-onset seizures, with or without secondary generalization.
3. Patients under titration phase (i.e., maintenance dose not reached yet according to clinical judgement) with cenobamate as adjunctive therapy in third or fourth line with 1 to maximum 2 (for third line)/3 (for fourth line) concomitant anti-seizure medications (ASMs).
4. Patients who have not been adequately controlled despite treatment with 2 or 3 (maximum) ASMs before cenobamate treatment initiation (including concomitant ASMs started before initiating cenobamate).
5. Patients with available retrospective data in medical charts, seizure diaries or patient's notes, including reliable information about seizure frequency (intended as the number of seizures and the corresponding time period) in the last 3 months before cenobamate treatment initiation.
6. Written informed consent (including consent for the processing of personal data) signed by the patient, or by the legally designated representative in case of patient lacking capacity, prior to entering the study following local regulation.

Exclusion Criteria:

1. Patients who meet any of the contraindications to the administration of cenobamate according to its approved Summary of Product Characteristics (SmPC).
2. Patients with progressive neurodegenerative central nervous system (CNS) diseases or (benign or malignant) brain tumors.
3. Patients with unstable psychiatric diagnosis, including suicidal ideation and behavior within 6 months prior to enrolment, current psychotic disorder, or acute mania.
4. Patients with known substance abuse or dependence (except for caffeine and nicotine).
5. Patients participating in any interventional study from cenobamate treatment initiation until enrolment visit.
6. Patients with ongoing pregnancy or breast-feeding from cenobamate treatment initiation until enrolment visit.
7. Patients who are seizure-free in the last 3 months before cenobamate treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by epilepsy with focal-onset seizures with or without secondary generalization who have not been adequately controlled despite a history of treatment with 2 or 3 anti-seizure medications (ASMs).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Responder rate | At 6 and at 12 months of maintenance treatment
  To describe the ≥50% responder rate during the 6 and 12 months of maintenance-dosing treatment with cenobamate with respect to the pretreatment baseline.

SECONDARY OUTCOMES:
Responder rate | At 6 and at 12 months of maintenance-dosing treatment
  To describe the ≥75%/≥90%/=100% responder rate during the 6 and 12 months of maintenance-dosing treatment with cenobamate with respect to the pre-treatment baseline.
Safety evaluation | 0 -12 months of maintenance-dosing treatment
  To describe real-world safety from treatment initiation until 12 months of maintenance-dosing treatment with cenobamate.
  Absolute and relative frequencies of patients treated with cenobamate who experienced at least one AE/Adverse Drug Reaction (ADR)/Serious Adverse Event (SAE)/Serious Adverse Drug Reaction (SADR)/AE of special interest during the observation period.
  Total number of AEs/ADRs/SAEs/SADRs/AEs of special interest occurred during the observation period.
Health-Related Quality of Life evaluation (QOLIE-31-P) | At 6 and at 12 months maintenance-dosing treatment
  QOLIE-31-P is a survey of health-related quality of life for adults with epilepsy. This questionnaire should be completed only by the person who has epilepsy (not a relative or friend). There are 39 questions about health and daily activities.The QOLIE-31-P consists of 38 self-reported items and is divided in eight parts which evaluate energy, mood, daily activities, cognition, medication effects, seizure worry, overall QoL , and health state. The first and the last items are scored with 0-10 and 0-100 scales, respectively, from the worst to the best situation. The remaining 36 items are scored using a Likert rating scale from 1 to 3,4,5, or 6. The raw scores are reorganized to have scores from 0 to 100. The final score is obtained from the subscale scores and is rescaled from 0 to 100 with higher scores associated with better QoL.
Health-Related Quality of Life evaluation (SF-6Dv2 ) | At 6 and at 12 months maintenance-dosing treatment
  The SF-6Dv2 Health Utility Survey provides keen insights into patient health and product performance by measuring six health domains.
  The SF-6Dv2™ Health Survey consists of six questions asking about different aspects of patient's health; for each question, patients should select the response (among 5 or 6 options per question) that best describe his/her health status.
Sleepiness status evaluation | At 6 and at 12 months of maintenance-dosing treatment
  To describe the sleepiness status of patients, by means of the Epworth Sleepiness Scale (ESS), at 6 and at 12 months of maintenance-dosing treatment with cenobamate.
  The ESS scale is designed to measure the patient's general level of daytime sleepiness.
  The ESS scale is designed to measure the patient's general level of daytime sleepiness and consists of 8 questions with a rating ranging from "0 = no chance of dozing" to "3 = high chance of dozing".
Healthcare resource evaluation | 0-12 months of maintenance-dosing treatment
  Absolute and relative frequencies of patients according to the type of resources used (ED accesses; inpatient hospitalizations; specialist outpatient visits; diagnostic exams) during the observation period.
  Descriptive statistics (mean, SD, median, 25th and 75th percentiles, min. and max.) of total number of resources used (ED accesses; inpatient hospitalizations; specialist outpatient visits; diagnostic exams) during the observation period.
  Descriptive statistics (mean, SD, median, 25th and 75th percentiles, min. and max.) of total duration of inpatient hospitalizations (calculated for each patient by summing the duration of all his/her inpatient hospitalizations) during the observation period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital TARNIER COCHIN, Paris, France, France